CLINICAL TRIAL: NCT03655431
Title: Telerehabilitation Using Kinect-based VR to Improve Mobility and Fatigue in Veterans With MS
Brief Title: Home Exercise Telerehabiliation for MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shane.Chanpimol (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Shane.Chanpimol, Co-Investigator, Washington D.C. Veterans Affairs Medical Center
Organization: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1846
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; rehabilitation; telerehabilitation; telehealth; veteran health; physical therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: An experimental and control group will be utilized. The experimental group will perform the telerehabilitation intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental): Physical therapists will develop an individualized program lasting 12 weeks depending on the needs of a given patient. Veterans will be seen 1 day/week via clinical video teleconferencing (CVT) for treatment. The rehabilitation protocol will last approximately 30 minutes with activities that are individualized to meet the participant's needs (range of motion, balance, strengthening, endurance, and functional activities). Patients assigned to telerehabilitation will utilize the VITAL rehab unit with Jintronix exercise package. Exercises, progression and rest periods will be administered and adjusted remotely by the physical therapist using a web-based clinical portal.
  Interventions: Other: Telerehabilitation; Other: Standard treatment

INTERVENTIONS:
Other: Telerehabilitation — Participants complete a standard physical therapy evaluation in-person. They are then provided telerehabilitation equipment for the telerehabilitation intervention. This intervention utilizes an Xbox Kinect sensor and tablet-based exercise software called Jintronix. The Jintronix exercise library includes an array of exercise activity options for varying functional levels. Exercise activities could be completed in sitting or standing postures and includes activities which focused on active range of motion, strength, balance, or calisthenic movements. Each activity requires the participant to complete a goal-directed game or replicate movements of an on-screen avatar. The therapist will adjust and progress the home exercise program using information provided by the Jintronix and the participant's verbal reports during clinical video teleconferencing. At the end of the intervention, the therapist will complete in-person discharge assessments.
Other: Standard treatment — Participants complete standard in-person physical therapy evaluation, follow-up, and treatment. Therapeutic exercise and activities will be prescribed to participants to perform at home between standard follow-up treatment appointments. At the end of the intervention, the physical therapist will complete in-person discharge assessments.

SUMMARY:
The primary purpose of this study is to evaluate the effects of an individualized telerehabilitation program on mobility, fatigue, and quality of life for Veterans with MS. The secondary purpose was to assess adherence to exercise recommendations and overall satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS based on the McDonald criteria
* Expanded Disability Status Scale (EDSS) of 3.0 - 6.5
* Cognitive ability (Montreal Cognitive Assessment score >23/30)
* Physician clearance for exercise participation
* Physical therapy referral

Exclusion Criteria:

* MS-related exacerbation within last 3 months
* Unstable cardiac or pulmonary disease
* Active substance abuse
* Uncontrolled seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Walking Scale-12 (MSWS-12) | Change after 12-week intervention
  This questionnaire has 12 items and measures self-reported walking ability in MS. The questions assess the limitations of a patient's walking due to MS during the past 2 weeks. Each item ranges from 1 to 5 and the higher the sum, the more severe the degree of limitation.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change after 12-week intervention
  The test involves assessments of clinician rated strength tests of standing balance, timed 3 meter walk, and five chair rise repetitions. The rating scale starts at "0" indicating no performance or low performance ranging to as score of "4" indicating high performance. The rating scale ranges from 0 to 12.
25-Foot Walk Test (25FWT) | Change after 12-week intervention
  The patient is instructed to walk 25 feet as fast as safely possible. Scoring the 25FW is the average of 2 trials that are performed consecutively. If necessary, assistive devices are allowed to be used.
Modified Fatigue Impact Scale (MFIS) | Change after 12-week intervention
  This is a standard measure used to measure fatigue. The scale consists of 21 items, with 10 items related to mental fatigue, and 11 items relating to physical and social fatigue. The scoring ranges between 0 and 82, a high score reflecting greater impact.
Veteran Rand 12 Quality of Life Measure (VR-12) | Change after 12-week intervention
  This 12-item questionnaire has eight principal physical and mental health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning, and mental health. The 12 items is summarized into two sub-scores measuring physical health and mental health.

OTHER OUTCOMES:
Patient Travel | Start of participation
  Patient reported estimates of commute to medical facility.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Wallin, MD, Principal Investigator — Washington DC VAMC
Locations (1):
- Washington DC VAMC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chanpimol S, Benson K, Maloni H, Conroy S, Wallin M. Acceptability and outcomes of an individualized exergaming telePT program for veterans with multiple sclerosis: a pilot study. Arch Physiother. 2020 Oct 1;10:18. doi: 10.1186/s40945-020-00089-5. eCollection 2020. PMID 33014426
- See also: Link to completed open-source publication. — https://archivesphysiotherapy.biomedcentral.com/articles/10.1186/s40945-020-00089-5